CLINICAL TRIAL: NCT04607603
Title: Efficacy of Cannabidiol in Treatment of Pain Due to Symptomatic Osteoarthritis of the Knee: A Randomized, Double-blind, Placebo-controlled Clinical Trial
Brief Title: Efficacy of Cannabidiol in Knee Osteoarthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Sibylle Pramhas, MD, Principal Investigator, Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Version 1.4
Record Dates: First submitted 2020-10-22; First posted 2020-10-29 (Actual); Last update posted 2022-10-05 (Actual); Status verified 2022-10

CONDITIONS: Osteo Arthritis Knee; Pain, Joint
MeSH Terms: conditions — Arthralgia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: double-blind placebo-controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cannabidiol (Experimental): In the Cannabidiol (CBD) arm CBD will be titrated up to 600 mg per die (titration 1 week) in capsules (3 daily doses) and maintained at 600mg per die (3 daily doses) for 7 weeks
  Interventions: Drug: Cannabidiol Oral Product
- Placebo (Placebo Comparator): In the placebo arm the placebo comparator will be administered in capsules in 3 daily doses
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cannabidiol Oral Product — Cannabidiol is administered in capsules. Each capsule contains 200mg of CBD administered 3 times daily to a total of 600mg per die
  Arms: Cannabidiol
Drug: Placebo — Placebo will be administered in capsules of identical appearance to CBD capsules in 3 doses per die
  Arms: Placebo

SUMMARY:
Painful symptomatic osteoarthritis (OA) of the knee is a very common disease, especially in older people (lifetime prevalence 9.5%). Current systemic pharmacological treatment options are limited.

Many patients presenting with knee osteoarthritis are of an advanced age and suffer from various co-morbidities. The benefit of the available systemic pharmacological treatment options in these patients can be summarized as uncertain. Therefore, the investigation of new symptomatic systemic pharmacological treatment options for knee OA is relevant. Even in patients without known contraindications, the treatment period with non-steroidal anti-inflammatory drugs should be kept short. It follows that the investigation of new potentially anti-inflammatory substances is of interest in symptomatic OA of the knee.

Cannabidiol has anti-inflammatory and analgesic properties in animal models. We therefore propose a randomised, double-blind, placebo-controlled clinical trial to investigate the potential efficacy of cannabidiol in painful symptomatic OA of the knee.

DETAILED DESCRIPTION:
Painful symptomatic osteoarthritis (OA) of the knee is a very common disease, especially in older people (lifetime prevalence 9.5%). Current systemic pharmacological treatment options are limited. The Osteoarthritis Research Society International recommends paracetamol, duloxetine, oral non-selective non-steroidal anti-inflammatory drugs and oral COX-2 inhibitors (anti-inflammatory substances) in patients without relevant concomitant diseases. In individuals with relevant concomitant diseases (diabetes, advanced age, high blood pressure, cardiovascular diseases, renal failure, gastrointestinal complications, depression, obesity), the recommendation for paracetamol, oral non-selective non-steroidal anti-inflammatory drugs and oral COX-2 inhibitors changes to 'inappropriate'.

In individuals with high co-morbidity risk (history of GI-bleeding, myocardial infarction, chronic renal failure) NSAIDs and oral COX-2 inhibitors are evaluated as inappropriate.

Many patients presenting with knee osteoarthritis are of an advanced age and suffer from various co-morbidities. The benefit of the available systemic pharmacological treatment options in these patients can be summarized as uncertain. Therefore, the investigation of new symptomatic systemic pharmacological treatment options for knee OA is relevant. Even in patients without known contraindications, the treatment period with non-steroidal anti-inflammatory drugs should be kept short. It follows that the investigation of new potentially anti-inflammatory substances is of interest in symptomatic OA of the knee.

Design

The planned study will be randomised, double-blind and placebo-controlled. 2 parallel groups will be investigated. One group will receive placebo, the other will receive 600mg cannabidiol per os during the treatment phase. The total study duration will be 13 weeks (2 weeks screening;

1 week titration phase; 7 weeks maintenance phase; 1 week tapering phase; 2 weeks follow-up) Main objective of the study will be to compare the change in the Western Ontario and McMasters Universities Osteoarthritis Index (WOMAC) Pain Index from baseline to the last week of the maintenance phase between the placebo and verum groups. The WOMAC Osteoarthritis Index is a validated patient questionnaire to assess symptoms and physical functional limitations in everyday life.

Secondary objectives include comparing the change in the WOMAC Function Index, the Global Patient Assessment of Gonarthrosis and the VAS Score. The planned number of participants is 86 (43 patients per group)

Measures/procedure After a 2-week screening phase, patients are randomised to a 1:1 placebo:verum after written consent. During the screening all patients are adjusted to a basic medication of 3 times 1g paracetamol/day. In the cannabidiol arm, titration is carried out within one week to the target dose of 600mg per day. This dosage is maintained for 7 weeks. This is followed by a balancing phase of 1 week. A follow-up is carried out 2 weeks after the maintenance phase is finished.

4 study visits are associated with blood sampling (safety laboratory) and physical examination and the completion of questionnaires and are carried out at our pain outpatient clinic. The remaining weekly visits are carried out by telephone.

During the entire duration of the study, patients are allowed the rescue medication of Tramadol 50mg up to 6/day.

ELIGIBILITY:
Inclusion Criteria:

Patient must be willing and able to give informed consent for participation in the study

* Age 18-80 years
* Knee Pain
* WOMAC Pain Subscale ≥ 5 during screening
* Fulfilment of the clinical criteria of the American College of Rheumatology for knee OA 13
* X-ray or MRI confirmation of knee osteoarthritis

All medications or interventions for pain due to knee osteoarthritis must have been stable for two weeks prior to screening and patient is willing to maintain a stable regimen throughout the study.

Exclusion Criteria:

Exclusion Criteria:

* Current mood disorder (dysthymia, bipolar mood disorder)
* Major Depression > 12 months (Beck Depression Inventory Score ≥ 18)
* History of a psychoactive substance use disorder within the preceding 12 months
* Major coexisting medical illness (e.g. severe heart failure, pulmonary hypertension, renal insufficiency)
* Glaucoma
* Acute myocardial infarction
* Uncontrolled hypertension
* History of convulsion
* Pregnancy; women of childbearing age will be required to use contraceptives during the duration of the study. Furthermore a pregnancy test will be performed prior to the beginning of the study and once a month during the study period.
* Breast feeding
* Participation in a clinical trial in the 3 weeks preceding the study
* Allergy to study medication
* Recent intra-articular corticosteroid or hyaluronic acid injection in the knee joint. Patients must be willing to abstain from such interventions during the entire study
* Use of the following medication:

  * opioids except for tramadol,
  * benzodiazepines other than indicated at low doses for sleep disorders
  * NSAID
  * Corticosteroids
* Impaired kidney function (Creatinine > 1.5mg/dl)
* Patient has significantly impaired hepatic function defined as any of the following:

  * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >5 × upper limit of normal (ULN).
  * ALT or AST >3 × ULN and (total bilirubin [TBL] >2 × ULN or international normalized ratio [INR] >1.5).
  * ALT or AST >3 × ULN with the presence of fatigue, nausea, vomiting, right upper quadrant pain or tenderness, fever, rash,and/or eosinophilia (>5%).
* Patient is currently using or has in the past used recreational or medicinal cannabis or synthetic cannabinoid based medications within 3 months prior to study entry
* Patient is unwilling to abstain from using recreational or medicinal cannabis, or synthetic cannabinoid based medications during the study
* Patients who are not able to understand the study measures and are not able to complete pain assessment forms.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2020-10-13 (Actual); Primary Completion 2022-02-17 (Actual); Study Completion 2022-03-29 (Actual)

PRIMARY OUTCOMES:
WOMAC Pain Score (WOMAC) Pain score | Change from baseline in WOMAC-Pain Index to the last week of the treatment phase (Week 8)
  Western Ontario and McMasters Universities Osteoarthritis Index (WOMAC) Pain Score Minimum=0 (best outcome) Maximum=10 (worst outcome)

SECONDARY OUTCOMES:
WOMAC Physical function | Change from baseline in WOMAC Physical function during the last week of the treatment phase (Week 8)
  Western Ontario and McMasters Universities Osteoarthritis Index (WOMAC) Physical function score Minimum=0 (best outcome) Maximum=10 (worst outcome)
Patient global assessment of Knee Osteoarthritis (PGA-KOA) | Change from baseline in PGA-KOA to PGA-KOA during the last week of the treatment phase (Week 8).
  PGA-KOA as compared to placebo
Use of Rescue Medication | Use of rescue mediaction during the 8 week treatment period
  Use of rescue medication in the placebo arm compared to the CBD Arm
Visual Analogue Scale (VAS) | Change mean 1 week VAS-Score from baseline to the last week of the treatment phase (Week 8)
  Mean VAS Score during 1 week as compared to placebo Minimum=0 (best outcome) Maximum=10 (worst outcome)
Health Related Quality of Life Score (SF-36) | Change of SF-36 score from baseline to the last week of the treatment phase (Week 8)
  Health Related Quality of Life Score (SF-36) as compared to placebo Minimum=0 (lowest level of health) Maximum=100 (highest level of health)
6 min walk-test | Change of 6 min walk test from baseline to the last week of the treatment phase (Week 8)
  6 min walk-test as compared to placebo
PainDETECT score | Change of PainDETECT score from baseline to the last week of the treatment phase (Week 8)
  PainDETECT score as compared to placebo Minimum= 0 (least likelihood neuropathic pain) Maximum=38 (highest likelihood neuropathic pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Medical University Vienna, Vienna, Austria

REFERENCES:
- [Derived] Pramhas S, Thalhammer T, Terner S, Pickelsberger D, Gleiss A, Sator S, Kress HG. Oral cannabidiol (CBD) as add-on to paracetamol for painful chronic osteoarthritis of the knee: a randomized, double-blind, placebo-controlled clinical trial. Lancet Reg Health Eur. 2023 Nov 10;35:100777. doi: 10.1016/j.lanepe.2023.100777. eCollection 2023 Dec. PMID 38033459